CLINICAL TRIAL: NCT04531722
Title: Intraoperative Brain Microdialysis to Assess Neuroinflammation in Epileptic Tissue Immediately Prior to Surgical Resection.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Charles L. Howe, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-000398
Record Dates: First submitted 2020-08-13; First posted 2020-08-28 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: We will establish intraoperative microdialysis in patients undergoing anterior temporal lobectomy for drug-resistant temporal lobe epilepsy. The human measurements will yield hypothesis-generating data and establish a methodological/logistical paradigm for future large-scale application of microdialysis in patients with drug refractory epilepsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- drug-resistant temporal lobe epilepsy (Experimental): Our current standard practice is to use a lateral approach through the middle temporal gyrus to place 3 depth electrodes targeting the hippocampus for intraoperative verification of pathological epileptiform activity prior to resection. Our research protocol will add one FDA approved electrode that has a central cannula for insertion of a microdialysis probe. The electro-physiological data that will be gathered is not altered and this methodology will not impact standard clinical care, except and will not to extend the duration in the OR - the measurements will occur during the clinical electrocorticography (ECoG; intracranial electroencephalography (iEEG)) procedure by 15 min.
  Interventions: Procedure: Intraoperative brain microdialysis

INTERVENTIONS:
Procedure: Intraoperative brain microdialysis — Our current standard practice is to use a lateral approach through the middle temporal gyrus to place 3 depth electrodes targeting the hippocampus for intraoperative verification of pathological epileptiform activity prior to resection. Our research protocol will add one FDA approved electrode that has a central cannula for insertion of a microdialysis probe.

SUMMARY:
This research study will investigate the fluid from the area of the brain that is being removed during clinical epilepsy surgery. The goal is to analyze this fluid for inflammatory markers that can potentially help identify new strategies in the future to control seizures in individuals with epilepsy who fail to respond to currently available drugs.

ELIGIBILITY:
Inclusion Criteria

* Failure to respond to at least two trials of anti-seizure drugs with different mechanisms of action
* Normal MRI

Exclusion Criteria

* Active immunomodulatory therapy
* Autoimmune disorder
* Signs or symptoms consistent with comorbid infection
* Oncological comorbidity

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Detection of analytes/protein | Through study completion, up to 5 years
  Presence of protein in the microdialysate

CONTACTS AND LOCATIONS:
Overall Officials: Charles Howe, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No